CLINICAL TRIAL: NCT07224815
Title: Development of a cfDNA 5mC/5hmC-based Epigenetic Biomarker Panel to Predict Chemotherapy Efficacy in Metastatic Colorectal Cancer
Brief Title: cfDNA 5mC/5hmC Biomarkers to Predict Chemotherapy Response in Metastatic Colorectal Cancer
Acronym: EpiCORE
Status: Recruiting | Type: Observational
Sponsor: City of Hope Medical Center (Other)
Responsible Party: Sponsor
Other Study IDs: 23228/EpiCORE
Record Dates: First submitted 2025-11-03; First posted 2025-11-05 (Actual); Last update posted 2025-11-05 (Actual); Status verified 2025-11

CONDITIONS: CRC (Colorectal Cancer)
Keywords: CRC; Colorectal cancer; 5mC; 5hmC; RAS/BRAF mutation; FOLFOX; FOLFIRI; hydroxymethylation
MeSH Terms: conditions — Colorectal Neoplasms

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (6):
- Discovery Cohort - PFS ≥ 12 Months (Responder): Patients with mCRC who achieved progression-free survival ≥ 12 months after first-line chemotherapy (FOLFOX or FOLFIRI).
  cfDNA 5mC/5hmC sequencing performed to identify epigenetic determinants of durable response.
  Interventions: Diagnostic Test: cfDNA 5mC/5hmC Sequencing (EpiCORE Discovery Phase)
- Discovery Cohort - PFS < 12 Months (Non-Responder): Patients with progression-free survival < 12 months after first-line chemotherapy.
  Compared with responders to identify epigenetic features associated with resistance.
  Interventions: Diagnostic Test: cfDNA 5mC/5hmC Sequencing (EpiCORE Discovery Phase)
- Training Cohort - PFS ≥ 12 Months (Responder): Independent mCRC cohort with long PFS (≥12M). Targeted sequencing (EpiCORE assay) to refine predictive markers.
  Interventions: Diagnostic Test: EpiCORE Assay (Targeted Sequencing / qPCR Validation)
- Training Cohort - PFS < 12 Months (Non-Responder): Independent mCRC cohort with short PFS (<12M). Targeted sequencing to validate resistance-associated markers.
  Interventions: Diagnostic Test: EpiCORE Assay (Targeted Sequencing / qPCR Validation)
- Validation Cohort - PFS ≥ 12 Months (Responder): Independent validation cohort analyzed with qPCR-based EpiCORE assay to confirm biomarker predictive accuracy.
  Interventions: Diagnostic Test: EpiCORE Assay (Targeted Sequencing / qPCR Validation)
- Validation Cohort - PFS < 12 Months (Non-Responder): Independent validation cohort with poor PFS analyzed to assess specificity and model performance.
  Interventions: Diagnostic Test: EpiCORE Assay (Targeted Sequencing / qPCR Validation)

INTERVENTIONS:
Diagnostic Test: cfDNA 5mC/5hmC Sequencing (EpiCORE Discovery Phase) — Genome-wide profiling of cfDNA methylation and hydroxymethylation from pre-treatment plasma to identify molecular determinants associated with chemotherapy efficacy (PFS ≥ 12M vs < 12M).
  Groups: Discovery Cohort - PFS < 12 Months (Non-Responder); Discovery Cohort - PFS ≥ 12 Months (Responder)
Diagnostic Test: EpiCORE Assay (Targeted Sequencing / qPCR Validation) — Targeted validation of cfDNA 5mC/5hmC markers from discovery phase using sequencing and qPCR to build and validate a predictive model for first-line chemotherapy response.
  Groups: Training Cohort - PFS < 12 Months (Non-Responder); Training Cohort - PFS ≥ 12 Months (Responder); Validation Cohort - PFS < 12 Months (Non-Responder); Validation Cohort - PFS ≥ 12 Months (Responder)

SUMMARY:
The EpiCORE study aims to identify cfDNA-based epigenetic markers predictive of response to first-line chemotherapy (FOLFOX or FOLFIRI) in metastatic colorectal cancer (mCRC).

By integrating 5-methylcytosine (5mC) and 5-hydroxymethylcytosine (5hmC) profiling, this study seeks to establish a non-invasive biomarker panel capable of distinguishing responders from non-responders.

DETAILED DESCRIPTION:
Despite the introduction of multi-agent chemotherapy regimens such as FOLFOX (5-FU, leucovorin, oxaliplatin) and FOLFIRI (5-FU, leucovorin, irinotecan), treatment outcomes in metastatic colorectal cancer (mCRC) remain highly variable.

Current predictive biomarkers, such as RAS/BRAF mutation or microsatellite instability, fail to accurately forecast response to cytotoxic chemotherapy.

Emerging evidence suggests that cfDNA methylation (5mC) and hydroxymethylation (5hmC) patterns reflect tumor biology and drug sensitivity, offering a promising avenue for precision chemotherapy.

The EpiCORE study integrates genome-wide 5mC/5hmC sequencing and targeted validation assays to identify and confirm epigenetic determinants of chemotherapy efficacy.

Discovery phase: Genome-wide 5mC/5hmC profiling of cfDNA from patients treated with first-line FOLFOX or FOLFIRI to identify candidate regions associated with treatment response.

Training phase: Targeted sequencing and model construction based on candidate loci.

Validation phase: qPCR-based testing to confirm predictive accuracy of the finalized EpiCORE panel.

This study aims to establish a robust cfDNA biomarker framework for predicting and monitoring chemotherapy response in mCRC, contributing to individualized therapeutic decision-making.

ELIGIBILITY:
Inclusion Criteria:

* Histologically confirmed metastatic colorectal adenocarcinoma (mCRC).
* Received first-line chemotherapy (FOLFOX or FOLFIRI).
* Availability of pre-treatment serum or plasma samples for cfDNA 5mC/5hmC analysis.
* Documented radiologic or clinical response evaluation (RECIST 1.1 or PFS-based).
* RAS/BRAF mutation status available.

Exclusion Criteria:

* Inadequate cfDNA yield or poor DNA quality.
* Non-adenocarcinoma histology.
* Active inflammatory or autoimmune disease that may alter cfDNA methylation.
* Concomitant malignancy requiring systemic therapy.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients diagnosed with Stage IV colorectal adenocarcinoma who received first-line FOLFOX or FOLFIRI chemotherapy and have available pre-treatment serum or plasma samples for cfDNA analysis.
Sampling Method: Non-Probability Sample
Enrollment: 600 (Estimated)
Dates: Start 2024-06-21 (Actual); Primary Completion 2026-06-18 (Estimated); Study Completion 2026-06-18 (Estimated)

PRIMARY OUTCOMES:
Progression-Free Survival (PFS) | Up to 36 months from initiation of first-line chemotherapy
  Progression-free survival (PFS) is defined as the time from initiation of first-line chemotherapy (FOLFOX or FOLFIRI) to the date of documented disease progression or death from any cause, whichever occurs first.
  The primary objective of the EpiCORE study is to evaluate whether cfDNA 5mC/5hmC-based biomarker profiles (EpiCORE panel) are associated with differences in PFS among patients with metastatic colorectal cancer (mCRC).

SECONDARY OUTCOMES:
Overall Survival (OS): | Up to 60 months from initiation of first-line chemotherapy
  Time from chemotherapy initiation to death from any cause

CONTACTS AND LOCATIONS:
Overall Officials: Ajay Goel, PhD, Principal Investigator — City of Hope Medical Center
Locations (1):
- City of Hope Medical Center, Duarte, California, United States

IPD SHARING:
Plan to Share IPD: No
Data collected for the study will be made available to others, including de-identified participant data, at publication, via a signed data access agreement and at the discretion of the investigators' approval of the proposed use of such data.

REFERENCES:
- [Background] Nelson MA, Shetty S, Kulakodlu M, Harley C, Seal B. A comparison of mortality and costs associated with FOLFOX versus FOLFIRI in stage IV colorectal cancer. J Med Econ. 2011;14(2):179-86. doi: 10.3111/13696998.2011.556693. Epub 2011 Feb 14. PMID 21319948
- [Background] Bond MJG, Bolhuis K, Loosveld OJL, de Groot JWB, Droogendijk H, Helgason HH, Hendriks MP, Klaase JM, Kazemier G, Liem MSL, Rijken AM, Verhoef C, de Wilt JHW, de Jong KP, Gerhards MF, van Amerongen MJ, Engelbrecht MRW, van Lienden KP, Molenaar IQ, de Valk B, Haberkorn BCM, Kerver ED, Erdkamp F, van Alphen RJ, Mathijssen-van Stein D, Komurcu A, Lopez-Yurda M, Swijnenburg RJ, Punt CJA; Dutch Colorectal Cancer Study Group. First-line systemic treatment strategies in patients with initially unresectable colorectal cancer liver metastases (CAIRO5): an open-label, multicentre, randomised, controlled, phase 3 study from the Dutch Colorectal Cancer Group. Lancet Oncol. 2023 Jul;24(7):757-771. doi: 10.1016/S1470-2045(23)00219-X. Epub 2023 Jun 14. PMID 37329889
- [Background] Bond MJG, Bolhuis K, Loosveld OJL, de Groot JWB, Droogendijk H, Helgason HH, Hendriks MP, Klaase JM, Kazemier G, Liem MSL, Rijken AM, Verhoef C, de Wilt JHW, de Jong KP, Gerhards MF, van Amerongen MJ, Engelbrecht MRW, van Lienden KP, Hermans JJ, Molenaar IQ, Grunhagen DJ, de Valk B, Haberkorn BCM, Kerver ED, Erdkamp F, van Alphen RJ, Mathijssen-van Stein D, Komurcu A, May AM, Swijnenburg RJ, Punt CJA; Dutch Colorectal Cancer Group. First-Line Systemic Treatment for Initially Unresectable Colorectal Liver Metastases: Post Hoc Analysis of the CAIRO5 Randomized Clinical Trial. JAMA Oncol. 2025 Jan 1;11(1):36-45. doi: 10.1001/jamaoncol.2024.5174. PMID 39570583
- [Background] Neugut AI, Lin A, Raab GT, Hillyer GC, Keller D, O'Neil DS, Accordino MK, Kiran RP, Wright J, Hershman DL. FOLFOX and FOLFIRI Use in Stage IV Colon Cancer: Analysis of SEER-Medicare Data. Clin Colorectal Cancer. 2019 Jun;18(2):133-140. doi: 10.1016/j.clcc.2019.01.005. Epub 2019 Jan 31. PMID 30878317
- [Background] Gibbons CE, Khan F. Dysphagia--a presenting symptom of forestier disease. J R Army Med Corps. 1996 Feb;142(1):32-3. doi: 10.1136/jramc-142-01-07. PMID 8667328
- [Background] Guler GD, Ning Y, Coruh C, Mognol GP, Phillips T, Nabiyouni M, Hazen K, Scott A, Volkmuth W, Levy S. Plasma cell-free DNA hydroxymethylation profiling reveals anti-PD-1 treatment response and resistance biology in non-small cell lung cancer. J Immunother Cancer. 2024 Jan 11;12(1):e008028. doi: 10.1136/jitc-2023-008028. PMID 38212123
- [Background] Ferrara R, Imbimbo M, Malouf R, Paget-Bailly S, Calais F, Marchal C, Westeel V. Single or combined immune checkpoint inhibitors compared to first-line platinum-based chemotherapy with or without bevacizumab for people with advanced non-small cell lung cancer. Cochrane Database Syst Rev. 2021 Apr 30;4(4):CD013257. doi: 10.1002/14651858.CD013257.pub3. PMID 33930176
- [Background] Baldassarre G, L de la Serna I, Vallette FM. Death-ision: the link between cellular resilience and cancer resistance to treatments. Mol Cancer. 2025 May 15;24(1):144. doi: 10.1186/s12943-025-02339-1. PMID 40375296
- [Background] Song D, Zhang Z, Zheng J, Zhang W, Cai J. 5-Hydroxymethylcytosine modifications in circulating cell-free DNA: frontiers of cancer detection, monitoring, and prognostic evaluation. Biomark Res. 2025 Mar 7;13(1):39. doi: 10.1186/s40364-025-00751-9. PMID 40055844
- [Background] Siegel RL, Kratzer TB, Giaquinto AN, Sung H, Jemal A. Cancer statistics, 2025. CA Cancer J Clin. 2025 Jan-Feb;75(1):10-45. doi: 10.3322/caac.21871. Epub 2025 Jan 16. PMID 39817679
- [Background] West-Szymanski DC, Zhang Z, Cui XL, Kowitwanich K, Gao L, Deng Z, Dougherty U, Williams C, Merkle S, Moore M, He C, Bissonnette M, Zhang W. Machine learning identifies cell-free DNA 5-hydroxymethylation biomarkers that detect occult colorectal cancer in PLCO Screening Trial subjects. bioRxiv [Preprint]. 2024 Feb 26:2024.02.25.581955. doi: 10.1101/2024.02.25.581955. PMID 38464122
- [Background] West-Szymanski DC, Zhang Z, Cui XL, Kowitwanich K, Gao L, Deng Z, Dougherty U, Williams C, Merkle S, He C, Zhang W, Bissonnette M. 5-Hydroxymethylated Biomarkers in Cell-Free DNA Predict Occult Colorectal Cancer up to 36 Months Before Diagnosis in the Prostate, Lung, Colorectal, and Ovarian Cancer Screening Trial. JCO Precis Oncol. 2024 Oct;8:e2400277. doi: 10.1200/PO.24.00277. Epub 2024 Oct 11. PMID 39393034
- [Background] Zeng C, Stroup EK, Zhang Z, Chiu BC, Zhang W. Towards precision medicine: advances in 5-hydroxymethylcytosine cancer biomarker discovery in liquid biopsy. Cancer Commun (Lond). 2019 Mar 29;39(1):12. doi: 10.1186/s40880-019-0356-x. PMID 30922396
- [Background] Xie YH, Chen YX, Fang JY. Comprehensive review of targeted therapy for colorectal cancer. Signal Transduct Target Ther. 2020 Mar 20;5(1):22. doi: 10.1038/s41392-020-0116-z. PMID 32296018
- [Background] Tirendi S, Marengo B, Domenicotti C, Bassi AM, Almonti V, Vernazza S. Colorectal cancer and therapy response: a focus on the main mechanisms involved. Front Oncol. 2023 Jul 19;13:1208140. doi: 10.3389/fonc.2023.1208140. eCollection 2023. PMID 37538108
- [Background] Koroukian SM, Booker BD, Vu L, Schumacher FR, Rose J, Cooper GS, Selfridge JE, Markt SC. Receipt of Targeted Therapy and Survival Outcomes in Patients With Metastatic Colorectal Cancer. JAMA Netw Open. 2023 Jan 3;6(1):e2250030. doi: 10.1001/jamanetworkopen.2022.50030. PMID 36656585
- [Background] Xu C, Mannucci A, Esposito F, Oliveres H, Alonso-Orduna V, Yubero A, Fernandez-Martos C, Salud A, Gallego J, Martin-Richard M, Fernandez-Plana J, Guillot M, Aparicio J, Fakih M, Kopetz S, Feliu J, Maurel J, Goel A. An Exosome-Based Liquid Biopsy Predicts Depth of Response and Survival Outcomes to Cetuximab and Panitumumab in Metastatic Colorectal Cancer: The EXONERATE Study. Clin Cancer Res. 2025 Mar 17;31(6):1002-1015. doi: 10.1158/1078-0432.CCR-24-1934. PMID 39820673